CLINICAL TRIAL: NCT04197895
Title: Clinical and Radiographic Evaluation of Advanced Platelet Rich Fibrin in the Preservation of Alveolar Ridge Following Atraumatic Tooth Extraction: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Advanced Platelet Rich Fibrin in the Preservation of Alveolar Ridge Following Atraumatic Tooth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nahed Gamal Saleh Abdelaal (Other)
Responsible Party: Sponsor-Investigator, Nahed Gamal Saleh Abdelaal, dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nana2019
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Socket Preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Socket preservation with APRF
  Interventions: Procedure: Socket preservation with APRF
- control group (Active Comparator): natural healing
  Interventions: Procedure: natural healing

INTERVENTIONS:
Procedure: Socket preservation with APRF — Socket preservation with APRF , A-PRF membranes were implanted into the extraction socket following tooth extraction. One entire A-PRF membrane would be placed at the base of the extraction socket and another A-PRF membrane will cover the extraction site then suturing will be done .Venous blood will be collected via venipuncture of the forearm with a butterfly needle into at least 10 mL sterile glass vacuum tube. The blood sample will be immediately centrifuged at 1,300 rpm (200 x g) for 8 minutes
  Arms: test group
Procedure: natural healing — after atraumatic extraction , the socket will be left for natural healing after suturing
  Arms: control group

SUMMARY:
compare the effect of application of A-PRF in socket preservation after atraumatic tooth extraction and natural healing regarding to bone remodeling . Null hypotheis, after atraumatic extraction, socket with advanced PRF has no difference with socket with blood clot in primary outcome

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are as follow :

  * patients with an unremarkable medical history
  * subjects with at least one site bordered by minimum of one tooth.
  * Nonsmoker
  * Teeth with root fracture, teeth with failed endodontic therapy or advanced caries
  * Intact extraction socket with no dehiscence or fenestration.
  * The buccolingual thickness of the buccal plate of bone in surgical area is 1 mm or more

Exclusion Criteria:

* Patients with systemic diseases.
* Patients with presence or history of osteonecrosis of the jaws, with use of bisphosphonates, exposure to head and neck radiation, chemotherapy.
* patients with large distinct pre-apical pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
mesial and distal height of extraction site | 2 months
  digital radiograph

SECONDARY OUTCOMES:
soft tissue thickness | 2 months
  will be evaluated by endo file with rubber stopper and digital caliper

IPD SHARING:
Plan to Share IPD: Undecided